CLINICAL TRIAL: NCT00584350
Title: Prevention of Contrast Nephropathy During Diagnostic Coronary Angiogram or PCI With Hydratation Based on LEVDP
Acronym: NEPHRON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Michel Nguyen, Doctor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 03-70-M5
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Radiographic Contrast Agent Nephropathy; Renal Failure; Coronary Heart Disease
Keywords: coronary angiogram; percutaneous coronary intervention
MeSH Terms: conditions — Renal Insufficiency; Coronary Disease | interventions — Sodium Bicarbonate; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: Hydratation according LVEDP + NaHCO3 (Experimental): Hydration with bolus of NaCl 0.9 to reach a LVEDP of 18 mmHg or more. This procedure is done while the patient is in the laboratory, with a catheter in the left ventricle.
  At the same time, an infusion of a sodium bicarbonate solution (150 mEq/L) is started at a rate of 1 ml/kg/h (max 110 ml/h) for 7 hours.
  Interventions: Other: Hydratation according LVEDP + NaHCO3
- B: Standard hydratation (Active Comparator): hydratation with normal saline (1 cc/kg/h; max 110 cc/h) starting at 8PM the day before the test and ending at 8PM the day of the test (24 hours total).
  Interventions: Other: normal saline
- C: Hydratation with sodium bicarbonate (Experimental): hydratation with sodium bicarbonate (150 mEq/L) at 3 cc/kg/h (max 330 cc/h) for 1 hour before the test and then, to be continued at 1 cc/kg/h (max 110 cc/h) for 6 hours (total of 7 hours of hydratation).
  Interventions: Other: Sodium bicarbonate

INTERVENTIONS:
Other: Hydratation according LVEDP + NaHCO3 — Hydration with bolus of NaCl 0.9 to reach a LVEDP of 18 mmHg or more. This procedure is done while the patient is in the laboratory, with a catheter in the left ventricle.
  At the same time, an infusion of a sodium bicarbonate solution (150 mEq/L) is started at a rate of 1 ml/kg/h (max 110 ml/h) for 7 hours.
  Arms: A: Hydratation according LVEDP + NaHCO3
Other: normal saline — hydratation with normal saline (1 cc/kg/h; max 110 cc/h) starting at 8PM the day before the test and ending at 8PM the day of the test (24 hours total).
  Arms: B: Standard hydratation
Other: Sodium bicarbonate — hydratation with sodium bicarbonate (150 mEq/L) at 3 cc/kg/h (max 330 cc/h) for 1 hour before the test and then, to be continued at 1 cc/kg/h (max 110 cc/h) for 6 hours (total of 7 hours of hydratation).
  Arms: C: Hydratation with sodium bicarbonate

SUMMARY:
The goal is to determine if prehydration based on LEVDP is superior to a standard hydratation with NaCl 0.9% or NaHCO3 for the prevention of contrast nephropathy related to a diagnostic coronary angiogram or to PCI.

DETAILED DESCRIPTION:
The goal is to determine if prehydration based on LEVDP is superior to a standard hydratation, independant of volemic status, with NaCl 0.9% or NaHCO3 for the prevention of contrast nephropathy related to a diagnostic coronary angiogram or to PCI.

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years old
* chronic renal insufficiency with a calculated creatinine clearance below 60 cc /min. (estimated with the MDRD formula)
* hemodynamically stable

Exclusion Criteria:

* Acute renal failure or in recuperation of acute renal failure
* urgent coronary angiogram
* moderate to severe valvulopathy or presence of a valvular prosthesis
* diagnostic of multiple myeloma
* dialysis before test
* having had a test with contrast product in the 2 weeks preceding
* receiving a nephrotoxic in the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2007-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of contrast nephropathy described as an increase of 44 micromol/L in plasma creatinine 48 hours after the injection of contrast product. | 48 hours

SECONDARY OUTCOMES:
changes in glomerular filtration in the 3 groups (measured with MDRD formula) | 48 hours
clinical events during the procedure or after (ex. pulmonary edema) | during hospitalisation
Incidence of contrast nephropathy defined as an increase of 25% of the creatinine value at 48 hours | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michel Nguyen, MD, FRCPC, Principal Investigator — Sherbrooke University
Locations (1):
- CHUS, clinical research center, Sherbrooke, Quebec, Canada